CLINICAL TRIAL: NCT06825845
Title: Long Term Follow-up Observational Study in Patients Treated with Gene-Modified T-Cell Therapy
Status: Not yet recruiting | Type: Observational
Sponsor: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CARs-LTFU-01
Record Dates: First submitted 2025-02-08; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Zevorcabtagene Autoleucel — Non-intervention

SUMMARY:
This is a prospective long-term follow-up (LTFU) study to evaluate the long-term safety and survival benefit for patients who received at least one of CARsgen's GM T cell product in a clinical trial or as a commercially available product. In this study, patients will be followed for up to 15 years after last GM T-cell infusion for the evaluation of delayed adverse events (AEs), vector persistence, potential risk for integration, and survival time due to GM T-cell exposure.

DETAILED DESCRIPTION:
As recommended by Health Authorities guidelines for human gene therapy products containing an integrated transgene, during the LTFU for 15 years after infusion, the information of the enrolled patients will be collected, including medical history, physical and laboratory-related examination data, AEs, survival information, etc. AEs recorded will include new malignancy, new or exacerbation infection, new or exacerbation neurological disease, new or exacerbation autoimmune disease etc. Samples will be obtained according to the schedule of activities, and laboratory tests will be conducted or preserved for future use.

All participants are recommended to be followed at least every six months for the first 5 years, and annually from the 6th year until at least 15 years or until informed consent withdrawal, loss to follow-up, or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

- 1. All patients who have received at least one GM T-cell infusion in the parent clinical study or in the post-approval setting.

2. Patients must be capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. For patients incapable of providing consent, the signed ICF of their legally accepted guardians must be obtained.

Exclusion Criteria:

* There are no specific exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Before any study procedure, informed consent must be signed by the participants, or by the participant's legal guardian for patients with no full civil capacity
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2039-12-31 (Estimated); Study Completion 2040-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess the risk of delayed AEs following exposure to GM T cells | 15 years

IPD SHARING:
Plan to Share IPD: No